CLINICAL TRIAL: NCT02802306
Title: Tack Optimized Drug Coated Balloon Angioplasty in the Superficial Femoral and Proximal Popliteal Arteries Using the Tack Endovascular System™
Brief Title: Tack Optimized Drug Coated Balloon Angioplasty Study of the Tack Endovascular System™ in Femoropoliteal Arteries
Acronym: TOBA III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA 0135
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Angioplasty; Peripheral Artery Disease; PAD; Lesion; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tack Implant (Experimental): Implantation of a Tack implant using the Intact Vascular Tack Endovascular System for the repair of post DCB-angioplasty dissections.
  Interventions: Device: Tack Endovascular System

INTERVENTIONS:
Device: Tack Endovascular System — Repair of post-PTA dissections using the Intact Vascular Tack Endovascular System
  Other Names: Post-PTA Dissection Repair Implant; Tack Implant; Tack Dissection Repair Device

SUMMARY:
This is an Outside the United States, post-CE Mark, multi-center, single-arm, non-blinded study designed to investigate the safety and efficacy of the Tack Endovascular System. This study will evaluate subjects with PAD who receive PTA (with a drug-coated balloon (DCB)) in the SFA and in popliteal arteries, ranging in diameter from 2.5mm to 6.0mm and lesion lengths of ≥20mm and ≤150mm, and have a resulting dissection(s) type(s) A through F. TOBA III will also evaluate the safety and efficacy of the device when used to treat a sub-group presenting with longer lesions of >150mm and ≤250mm.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all of the following inclusion criteria to be eligible for enrollment:

  1. Male or non-pregnant Female ≥ 18 years of age at the time of consent
  2. Female subjects of childbearing potential must have a negative pregnancy test prior to treatment and must use some form of contraception through the duration of the study
  3. Target limb requires no additional treatment aside from the target lesion and the iliac artery(ies) during the index procedure
  4. Subject or has been informed of and understands the nature of the study and provides signed informed consent to participate in the study. If the subject possesses the ability to understand and provide informed consent but due to physical inability, the subject cannot sign the ICF, an impartial witness may sign on behalf of the subject
  5. Willing to comply with all required follow-up visits
  6. Rutherford Classification 2, 3 or 4
  7. Estimated life expectancy >1 year
  8. Eligible for standard surgical repair, if necessary
  9. Subject is ambulatory (assistive devices such as a cane or walker is acceptable

Exclusion Criteria:

* Subject must NOT meet any of the following exclusion criteria to be eligible for enrollment:

  1. Rutherford Classification 0, 1, 5 or 6
  2. Is pregnant or refuses to use contraception through the duration of the study
  3. Previous infrainguinal bypass graft in the target limb
  4. Planned amputation on the target limb
  5. Systemic infection or infection within the target limb and/or immunocompromised
  6. Endovascular or surgical procedure (not including diagnostic procedures) on the target limb within 30 days prior to or within 30 days after the index procedure
  7. Endovascular or surgical procedure (not including diagnostic procedures) on the non-target limb within 14 days prior to the index procedure or planned procedure within 30 days after the index procedure
  8. Prior coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) procedure within 30 days prior to the index procedure or planned CABG/PCI within 30 days after the index procedure
  9. Any other previous or planned surgical or endovascular procedure (not including diagnostic procedures) within 14 days prior to or 30 days post index procedure
  10. Planned atherectomy, cryoplasty, stenting or any other treatment (with the exception of a crossing device) of the target lesion other than PTA during the index procedure
  11. Known coagulopathy, hypercoagulable state, bleeding diathesis, other blood disorder, or a platelet count less than 80,000/microliter or greater than 500,000/microliter
  12. Known hypersensitivity or allergy to antiplatelet or anticoagulant therapy
  13. Myocardial infarction within 30 days prior to enrollment
  14. History of stroke within 90 days prior to enrollment
  15. Serum creatinine of >2.5 mg/dL
  16. Requires treatment of tibial or outflow vessels at the index procedure, which include the P2 and P3 segments of the popliteal artery and the tibioperoneal vessels
  17. Known hypersensitivity or contraindication to nickel-titanium alloy (Nitinol)
  18. Participating in another ongoing investigational clinical trial that has not completed its primary endpoint
  19. Has other comorbidities that, in the opinion of the investigator, would preclude them from receiving this treatment and/or participating in study-required follow-up assessments
  20. Known hypersensitivity or allergy to contrast agents that cannot be medically managed
  21. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-06; Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Safety - Freedom from the occurrence of any new-onset major adverse event(s) | 30 days
  Freedom from the occurrence of any new-onset major adverse event(s) (MAEs) defined as index limb amputation (above the ankle), CEC adjudicated clinically-driven target lesion revascularization (CD-TLR), or all-cause death at 30 days.
Efficacy - Primary Patency | 12 months
  Primary patency defined as freedom from CEC adjudicated clinically driven target lesion revascularization (CD-TLR) and freedom from core lab adjudicated duplex ultrasound derived binary restenosis at 12 months (defined as PSVR >2.5:1).

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, MD, Principal Investigator — Medical University Hospital Graz
Locations (17):
- University Hospital AKH Vienna, Vienna, Austria
- Belgium (2):
  - Imelda Hosptial, Bonheiden
  - A.Z. St. Blasius Hospital, Dendermonde
- Germany (12):
  - Karolinen-Hospital Klinik für Angiologie Arnsberg Clinic, Arnsberg
  - Universitats-Herzzentrum Freiburg-Bad Krozingen Klinik fur Kardiologie und Angiologie lI, Bad Krozingen
  - Franziskus-Hospital Berlin, Berlin
  - Medizinische Klinik II Fürst Stirum Klinik Bruchsal, Bruchsal
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Asklepios Klinik St. Georg Herz-, Gefäß- und Therapiezentrum, Abt. Klinische und Interventionelle Angiologie, Hamburg
  - Center for Cardiology & Vascular Intervention, Hamburg
  - Westküstenklinikum Heide, Heide
  - Herz und Gefäßzentrum im Klinikverbund Oberallgäu-Kempten, Immenstadt im Allgäu
  - Klinikum Karlsbad Langensteinbach, Karlsbad
  - Universitätsklinik Leipzig, Leipzig
  - Universitätsmedizin Mainz II Medizinische Klinik und Poliklinik, Angiologie, Mainz
- Switzerland (2):
  - Cantonal Hospital Lucerne Division of Angiology, Lucerne
  - Ospedale Regionale di Lugano - Civico e Italiana Civico, Lugano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brodmann M, Wissgott C, Brechtel K, Nikol S, Zeller T, Lichtenberg M, Blessing E, Gray W; TOBA III Investigators. Optimized drug-coated balloon angioplasty of the superficial femoral and proximal popliteal arteries using the Tack Endovascular System: TOBA III 12-month results. J Vasc Surg. 2020 Nov;72(5):1636-1647.e1. doi: 10.1016/j.jvs.2020.01.078. Epub 2020 May 12. PMID 32414527